CLINICAL TRIAL: NCT00006354
Title: Phase I Clinical Trial of Recombinant Viscumin (rViscumin, rMistletoe Lectin, rML) Administered Twice Weekly By The Intravenous Route In Patients With Solid Tumors After Failure of Standard Therapy
Brief Title: Mistletoe Lectin in Treating Patients With Advanced Solid Tumors That Have Not Responded to Previous Therapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: EORTC-16002; EORTC-16002
Record Dates: First submitted 2000-10-04; First posted 2003-01-27 (Estimated); Last update posted 2012-07-24 (Estimated); Status verified 2012-07

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific

INTERVENTIONS:
Dietary Supplement: mistletoe extract

SUMMARY:
RATIONALE: Mistletoe lectin may slow the growth of cancer cells and be an effective treatment for solid tumors.

PURPOSE: Phase I trial to study the effectiveness of mistletoe lectin in treating patients who have advanced solid tumors that have not responded to previous therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose and dose-limiting toxicity of mistletoe lectin (recombinant viscumin) in patients with advanced solid tumors who have failed standard therapy.
* Determine the pharmacokinetics of this regimen in these patients.
* Determine whether induction of antibodies against recombinant viscumin occurs in these patients.
* Determine whether immunological stimulation at the RNA level of immune cells occurs in patients treated with this regimen.
* Determine whether modification of endothelial parameters occurs in patients treated with this regimen.
* Determine the objective response rates in patients treated with this regimen.

OUTLINE: This is a dose-escalation study.

Patients receive mistletoe lectin (recombinant viscumin) IV over 1 hour twice weekly. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.

Cohorts of 1-3 patients receive escalating doses of recombinant viscumin until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which 20% of patients experience dose-limiting toxicity during the first course. Additional patients are treated at the MTD.

Patients are followed every 3 months until disease progression or initiation of another therapy.

PROJECTED ACCRUAL: A minimum of 37 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically proven progressive advanced solid tumor that is not amenable to standard therapy (i.e., resistant to standard therapy or for which no standard therapy exists)
* No clinically symptomatic CNS involvement

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* At least 3 months

Hematopoietic:

* WBC at least 3,000/mm^3
* Neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* AST and ALT less than 2.5 times ULN (5 times ULN if liver metastases present)
* Alkaline phosphatase less than 2.5 times ULN (5 times ULN if liver metastases present)

Renal:

* Creatinine less than 1.4 mg/dL

Cardiovascular:

* No ECG abnormalities of clinical relevance

Other:

* No severe or unstable systemic disease or infection
* No circumstances (e.g., alcoholism or substance abuse) that would preclude study participation
* HIV negative
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 4 weeks since prior immunostimulating substances, biologic response modifiers, or colony-stimulating factors
* No concurrent immunostimulating substances, colony-stimulating factors (except in life-threatening situations), biologic response modifiers, or monoclonal antibodies

Chemotherapy:

* At least 4 weeks since prior chemotherapy

Endocrine therapy:

* At least 4 weeks since prior hormonal therapy
* At least 4 weeks since prior systemic steroids
* No concurrent systemic steroids

Radiotherapy:

* At least 4 weeks since prior radiotherapy
* No concurrent radiotherapy

Surgery:

* Not specified

Other:

* No prior mistletoe preparations
* At least 4 weeks since prior investigational treatment
* No other concurrent anticancer agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2000-08; Primary Completion 2003-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Schoffski, MD, MPH, Study Chair — Hannover Medical School
Locations (2):
- Centre Regional Rene Gauducheau, Nantes-Saint Herblain, France
- Medizinische Hochschule Hannover, Hanover, Germany